CLINICAL TRIAL: NCT00346515
Title: Evaluating the Use of the FiberNet® Emboli Protection Device in Carotid Artery Stenting: The EPIC US Feasibility Study
Brief Title: EPIC US Feasibility Study: Use of the FiberNet® Emboli Protection Device in Carotid Artery Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumen Biomedical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 864
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery; carotid stenosis; carotid stenting; embolic protection
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: FiberNet Emboli Protection System

SUMMARY:
Multicenter, prospective, feasibility study designed to demonstrate the performance and safety of the Lumen Biomedical, Inc. FiberNet™ Embolic Protection System as an adjunctive device during carotid artery percutaneous intervention using the Guidant Acculink carotid stent in high surgical risk patients.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the high surgical risk criteria.
* Candidate for percutaneous stenting with target lesion located within common or internal carotid artery.
* Symptomatic with atherosclerotic stenosis ≥ 50% or asymptomatic with atherosclerotic stenosis ≥ 70% of the carotid artery by NASCET Criteria.

Exclusion Criteria:

* Allergy to Heparin.
* Myocardial infarction within the last 14 days.
* Angioplasty or PTCA/PTA procedure within the past 48 hours.
* Cardiac surgery within the past 60 days.
* Planned invasive surgical procedure within 30 days.
* Stroke within the past 14 days.
* Transient ischemic neurological attack (TIA) or amaurosis fugax within the past 48 hours.
* Intracranial stenosis that exceeded the severity of an extracranial stenosis.
* Peripheral vascular disease of sufficient severity to prevent vascular access to the target lesion.
* Total occlusion of the target vessel.
* Lesion within 2cm of the ostium of the common carotid artery.
* A stenosis that is known to be unsuitable for stenting because of one or more of:

  1. Tortuous or calcified anatomy proximal or distal to the stenosis
  2. Presence of visual thrombus
  3. Pseudo occlusion ('string sign')
* Serial lesions that requires more then one stent to cover entire lesion.
* Procedural complication prior to introduction of the FiberNet device into the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-06; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The rate of all death, all stroke and myocardial infarction within 30 days of the procedure.

SECONDARY OUTCOMES:
All death and all stroke rates; Non-stroke neurological event rates; Technical success rates; Procedural success rates; Access site complication rates

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Bacharach, MD, Principal Investigator — North Central Heart Institute
Locations (4):
- United States (4):
  - Hoag Hospital, Newport Beach, California
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Riverside Methodist Hospital, Columbus, Ohio
  - North Central Heart Institue, Sioux Falls, South Dakota